CLINICAL TRIAL: NCT07295119
Title: Randomized Interventional Clinical Trial Involving Patient Undergoing Cataract Surgery Aiming To Evaluate The Halo Perception After Implantation Of Extended Depth Of Focus Intraocular Lenses (IOLs) Compared To Trifocal IOLs
Brief Title: Evaluation Of Patient Satisfaction And Quality Of Vision After EDOF Or Trifocal IOL Implantation
Acronym: TRIEDOF IOLS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Principal Investigator, Emilio Pedrotti, Full Professor of Ophthalmology and Chairman Director, School of Ophthalmology Eye Clinic - Department of Surgery, Dentistry, Pediatrics and Gynecology, Azienda Ospedaliera Universitaria Integrata Verona
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 74253-12/12/2022
Record Dates: First submitted 2025-12-03; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Cataract; Presbyopia Correction
Keywords: EDOF IOL; Trifocal IOL; Halo perception; spectacle indipendente
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Intervention Model Description: This is a two-arm, parallel-group, randomized clinical study in which each participant receives bilateral cataract surgery followed by implantation of prespecified intraocular lenses (IOLs) according to group assignment. Participants in the experimental arm receive a mixed-modality approach using two different EDOF IOL models implanted contralaterally, while participants in the control arm receive bilateral implantation of the same trifocal IOL model. Randomization occurs at the participant level, and both eyes follow the allocated intervention strategy. All assessments and follow-up visits proceed in parallel for both groups using standardized procedures.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants are masked to the intraocular lens (IOL) model implanted in each eye. Outcome assessors, including performing postoperative visual testing and halometry, remain masked to treatment allocation. Surgical staff cannot be masked due to required knowledge of lens type during the procedure. Postoperative data collection is structured to prevent assessors from accessing operative records or lens identifiers. Patients are instructed not to discuss perceived optical differences between eyes during masked assessments to preserve masking integrity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fusion EDOF IOL (Experimental): Participants undergo bilateral cataract surgery with contralateral implantation of two different extended-depth-of-focus intraocular lenses. The Mini Well IOL is implanted in the dominant eye and the Mini Well Proxa IOL in the non-dominant eye. This combined optical strategy is intended to provide continuous functional vision across distances while potentially reducing dysphotopsia by leveraging complementary lens designs. All procedures follow standardized surgical and postoperative protocols.
  Interventions: Device: Fusion EDOF IOL Implantation
- Bilateral Trifocal IOL (Active Comparator): Participants undergo bilateral cataract surgery with implantation of the same trifocal intraocular lens, the FineVision POD F, in both eyes. The lens distributes light across distance, intermediate, and near focal points and represents a standard presbyopia-correcting approach. Surgical technique and postoperative management are consistent with those used in the experimental arm to ensure comparability.
  Interventions: Device: Bilateral Trifocal IOL Implantation

INTERVENTIONS:
Device: Fusion EDOF IOL Implantation — Bilateral cataract extraction followed by implantation of two different extended-depth-of-focus intraocular lenses in opposite eyes. The dominant eye receives an EDOF lens based on wavefront-modulation optics (Mini Well), while the non-dominant eye receives a complementary EDOF lens optimized for near to intermediate performance (Mini Well Proxa). This contralateral design is intended to extend functional vision range and modulate dysphotopsia by combining distinct optical profiles within the same participant.
  Arms: Fusion EDOF IOL
Device: Bilateral Trifocal IOL Implantation — Bilateral cataract extraction followed by implantation of the same trifocal presbyopia-correcting intraocular lens in both eyes (FineVision POD F). This lens allocates light across three focal points-distance, intermediate, and near-representing a standard multifocal approa
  Arms: Bilateral Trifocal IOL

SUMMARY:
Brief Summary of the Study

The goal of this clinical study is to compare the quality of vision and patient satisfaction after cataract surgery using two different approaches to multifocal intraocular lenses (IOLs). These lenses replace the natural lens removed during surgery and are designed to allow clear vision at near, intermediate, and far distances, reducing or eliminating the need for glasses.

The study aims to understand whether using two different lens models-Mini Well in the dominant eye and Mini Well Proxa in the non-dominant eye-produces different levels of visual quality, glare, halos, or overall satisfaction compared with implanting the same trifocal lens model (FineVision POD F) in both eyes.

All lenses included in the study are approved medical devices already available on the market.

Who can participate? Adults scheduled to undergo cataract surgery in both eyes at the Ophthalmology Unit of the Policlinico of Verona may be eligible. A total of 36 participants will take part.

How does the study work?

Participation is voluntary. After informed consent, participants are randomly assigned (like flipping a coin) to one of two groups:

1. Experimental group: Mini Well lens in the dominant eye and Mini Well Proxa lens in the other eye.
2. Comparison group: FineVision POD F lens in both eyes.

Neither participants nor the clinical team conducting postoperative assessments will know which lenses were implanted (blinded study).

Before surgery, participants undergo a standard ophthalmic evaluation, including visual acuity tests and measurements of eye structure. After surgery in each eye, follow-up visits take place at approximately 1-2 days, 14 days, 1 month, and 3 months. During these visits, clinicians assess visual performance, eye health, and any symptoms. At the 3-month visit, participants also complete a questionnaire on vision quality and satisfaction, and undergo a specific test to measure perception of halos.

Participant responsibilities Participants are asked to attend all scheduled visits, follow medical instructions, use prescribed medications, and promptly report any symptoms or concerns.

Potential benefits Participants may experience improved vision at all distances with reduced dependence on glasses. However, personal benefit cannot be guaranteed. The study is expected to help determine whether combining two different lens models provides better visual outcomes than using the same lens in both eyes.

Risks and discomforts Risks are the same as those associated with standard cataract surgery and multifocal IOLs, including rare surgical complications and the possibility of visual disturbances such as glare or halos. These symptoms are common with multifocal lenses and often diminish over time, but in rare cases may require further intervention. All adverse events will be closely monitored.

Alternatives Patients may choose standard cataract surgery with monofocal lenses, which usually provide clear vision at one distance and may still require glasses for intermediate or near vision. Declining participation will not affect the quality of care.

Duration Each participant's involvement lasts about 4 months.

Voluntary participation Participants may withdraw at any time without affecting their medical care.

Confidentiality All personal and medical information will be handled confidentially and used only according to privacy regulations. Study results may be published anonymously in scientific reports.

DETAILED DESCRIPTION:
This study is designed to evaluate patient-reported satisfaction and visual quality following bilateral cataract surgery with implantation of two different multifocal intraocular lens (IOL) strategies. The investigation compares a mixed-modality combination of complementary extended-depth-of-focus (EDOF) IOLs with a bilateral trifocal IOL approach. Although all lenses included in this research are CE-marked and commercially available, they differ in optical architecture and light-distribution profiles, offering an opportunity to assess whether pairing distinct optical designs between eyes can mitigate dysphotopsia while maintaining a full range of functional vision.

The scientific rationale derives from the known trade-offs associated with presbyopia-correcting IOLs. Trifocal designs distribute light to three focal points and provide distance, intermediate, and near performance, but may also induce photic phenomena such as halos or glare. EDOF platforms extend the depth of focus through controlled modulation of spherical aberration or wavefront shaping, with the goal of improving image continuity and contrast. The Mini Well and Mini Well Proxa lenses, which incorporate different wavefront-engineering profiles, are hypothesized to act synergistically when implanted contralaterally. This design may reduce dysphotopsia intensity by balancing light distribution asymmetrically across the visual system. In contrast, bilateral FineVision POD F implantation represents a uniform, widely adopted trifocal strategy.

The study is conducted at the Ophthalmology Unit of the Policlinico of Verona and enrolls 36 patients requiring routine bilateral cataract extraction. Participants are randomized 1:1 to one of the two treatment groups. The allocation sequence is computer-generated and concealed using a predefined method to ensure unbiased assignment. Masking is maintained at the patient level; patients are not informed of the IOL type they receive. Outcome assessors remain masked whenever feasible, although surgeons cannot be masked due to the nature of the intervention.

The protocol follows a standardized clinical workflow. Preoperative evaluation includes refraction, slit-lamp biomicroscopy, tonometry, retinal assessment, and biometric measurements using optical biometry to calculate IOL power. Cataract extraction is performed using a uniform phacoemulsification technique, with efforts to standardize incision size and capsulorhexis configuration. Postoperative care follows standard clinical practice and includes scheduled visits at early, intermediate, and late postoperative time points for both eyes.

Across follow-up, participants undergo routine ophthalmic assessments and standardized testing. At the final postoperative visit, patients complete structured questionnaires addressing visual function, satisfaction, spectacle independence, and visual disturbances. Objective quantification of dysphotopsia, including halo intensity and size, is also performed using validated halometry tools. These assessments provide combined subjective and objective characterization of visual quality.

The anticipated duration of participation is approximately four months, including preoperative evaluation, surgery for each eye, and postoperative follow-up through the three-month visit after the second eye procedure. Study data are collected in case report forms and stored under coded identifiers to ensure confidentiality. Data management follows applicable privacy legislation and good clinical practice guidelines. Quality assurance procedures include verification of source documents, consistency checks for questionnaire scoring, and calibration of devices used for optical quality measurements.

By comparing a contralateral EDOF-based strategy with bilateral trifocal implantation, this investigation seeks to clarify whether mixing complementary optical designs yields advantages in patient satisfaction, visual comfort, or dysphotopsia reduction. The findings are expected to contribute evidence relevant to presbyopia-correcting IOL selection, optimization of binocular optical planning, and patient counseling in cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Diagnosis of age-related cataract in both eyes requiring bilateral cataract surgery.
* Corneal astigmatism 0.50 diopters or less in each eye.
* No other media opacities except cataract.
* Regular corneal shape without abnormal curvature or high-order aberrations on topography/aberrometry.
* Intraocular lens spherical power between +10.00 and +30.00 diopters according to biometry and IOL calculation.
* Willing and able to undergo surgery in the second eye within 7 days of the first-eye surgery.
* Willing and able to attend all scheduled follow-up visits, including the 3-month visit.
* Able to understand the study information and provide written informed consent.

Exclusion Criteria:

* Any prior ocular surgery in either eye.
* Any concomitant ocular disease that could affect visual outcomes (for example glaucoma, retinal disease, significant macular pathology, corneal dystrophy or degeneration, keratoconus, significant dry eye not controlled with treatment).
* Clinically significant irregular astigmatism or corneal scarring.
* Any intraoperative complication during cataract surgery that could compromise IOL position or visual outcome (such as posterior capsule rupture, zonular dialysis); such eyes will be excluded from the analysis set.
* Significant posterior capsule opacification before the 3-month outcome visit requiring YAG capsulotomy.
* Systemic disease or neurological condition that, in the investigator's opinion, may affect visual function, ability to complete testing (for example halometry, questionnaires), or study participation.
* Cognitive impairment or psychiatric condition that precludes giving informed consent or complying with study procedures.
* Participation in another interventional clinical study that could interfere with outcomes of this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-04-24 (Actual); Primary Completion 2024-11-13 (Actual); Study Completion 2024-11-13 (Actual)

PRIMARY OUTCOMES:
Objective halo area under binocular vision. | 3 months post-second eye surgery.
  Objective halo area under binocular vision, defined as the quantitative measurement of halo perception expressed as the total area (cm²) of the halo pattern surrounding a central light stimulus under binocular conditions, assessed 3 months after bilateral intraocular lens (IOL) implantation (3 months post-second eye surgery). Higher halo area values indicate more pronounced photic phenomena (worse halo disturbance), whereas lower values indicate fewer or less extensive halos (better outcome)

SECONDARY OUTCOMES:
Uncorrected Distance Visual Acuity (UDVA) | 1 and 3 months postoperatively.
  Monocular and binocular uncorrected distance visual acuity (UDVA) at 4 m, measured in logarithm of the minimum angle of resolution (logMAR) units, assessed at 1 and 3 months postoperatively. The logMAR scale has lower values indicating better visual acuity, with 0.0 logMAR corresponding to 20/20 Snellen-equivalent vision and negative values representing better than 20/20.
Uncorrected Intermediate Visual Acuity (UIVA) | 1 and 3 months postoperatively.
  Monocular and binocular uncorrected intermediate visual acuity (UIVA) at 80 cm, measured in logarithm of the minimum angle of resolution (logMAR) units, assessed at 1 and 3 months postoperatively. The logMAR scale has lower values indicating better visual acuity, with 0.0 logMAR corresponding to 20/20 Snellen-equivalent vision and negative values representing better than 20/20.
Uncorrected Near Visual Acuity (UNVA) | 3 months postoperatively.
  Monocular and binocular uncorrected near visual acuity (UNVA) at 40 cm, measured in logarithm of the minimum angle of resolution (logMAR) units, assessed 3 months postoperatively. The logMAR scale has lower values indicating better visual acuity, with 0.0 logMAR corresponding to 20/20 Snellen-equivalent vision and negative values representing better than 20/20.
Contrast Sensitivity (CS) | 3 months postoperatively.
  Binocular contrast sensitivity measured with the CSV-1000 under photopic and scotopic conditions at spatial frequencies of 3, 6, 12, and 18 cycles per degree (cpd), assessed 3 months postoperatively. Contrast sensitivity is reported in log units for each spatial frequency, with higher values indicating better visual performance (greater ability to detect low-contrast targets).
Strehl Ratio | 3 months postoperatively
  Strehl ratio of the total eye measured with the OSIRIS-T aberrometer at a 4 mm pupil diameter, 3 months postoperatively. The Strehl ratio is a dimensionless index of optical quality ranging from 0 to 1, with values closer to 1 indicating better optical quality and less optical degradation
Root Mean Square | 3 months postoperatively
  Root Mean Square (RMS) higher-order aberration (µm) of the total eye measured with the OSIRIS-T aberrometer at a 4 mm pupil diameter, 3 months postoperatively. Lower RMS values indicate fewer aberrations and thus a better optical outcome; there is no fixed minimum or maximum, but values in healthy eyes are typically in the submicrometer range.
Quality of Life (NEI RQL-42 Score) | 3 months postoperatively
  Patient-reported satisfaction assessed using the National Eye Institute Refractive Error Quality of Life-42 (NEI-RQL-42) questionnaire at 3 months postoperatively. The NEI-RQL-42 provides multi-domain scores transformed to a 0-100 scale, with higher scores indicating better refractive error-related quality of life and greater satisfaction with vision.

CONTACTS AND LOCATIONS:
Locations (1):
- AOUI Verona, Verona, Verona, Italy

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data that underlie the main published results (including primary and secondary outcomes) will be shared. Data will be available beginning 12 months after publication of the primary manuscript and for 5 years thereafter. Data will be shared with qualified researchers for methods-sound proposals focused on cataract surgery, intraocular lenses, or visual outcomes, after approval by the sponsor and execution of a data use agreement. Requests should be sent to the corresponding investigator by email.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data will be available beginning 12 months after publication of the primary manuscript and for 5 years thereafter.
Access Criteria: Data will be shared with qualified researchers for methods-sound proposals focused on cataract surgery, intraocular lenses, or visual outcomes, after approval by the sponsor and execution of a data use agreement. Requests should be sent to the corresponding investigator by email.

REFERENCES:
- [Background] Pedrotti E, Neri E, Bonacci E, Barosco G, Galzignato A, Montresor A, Rodella A, De Gregorio A, Bosello F, Marchini G. Extended Depth of Focus Versus Monofocal IOLs in Patients With High Myopia: Objective and Subjective Visual Outcomes. J Refract Surg. 2022 Mar;38(3):158-166. doi: 10.3928/1081597X-20211220-01. Epub 2022 Mar 1. PMID 35275002
- [Background] Pedrotti E, Chierego C, Talli PM, Selvi F, Galzignato A, Neri E, Barosco G, Montresor A, Rodella A, Marchini G. Extended Depth of Focus Versus Monofocal IOLs: Objective and Subjective Visual Outcomes. J Refract Surg. 2020 Apr 1;36(4):214-222. doi: 10.3928/1081597X-20200212-01. PMID 32267951
- [Background] de Medeiros AL, de Araujo Rolim AG, Motta AFP, Ventura BV, Vilar C, Chaves MAPD, Carricondo PC, Hida WT. Comparison of visual outcomes after bilateral implantation of a diffractive trifocal intraocular lens and blended implantation of an extended depth of focus intraocular lens with a diffractive bifocal intraocular lens. Clin Ophthalmol. 2017 Oct 26;11:1911-1916. doi: 10.2147/OPTH.S145945. eCollection 2017. PMID 29138533
- [Background] Khandelwal SS, Jun JJ, Mak S, Booth MS, Shekelle PG. Effectiveness of multifocal and monofocal intraocular lenses for cataract surgery and lens replacement: a systematic review and meta-analysis. Graefes Arch Clin Exp Ophthalmol. 2019 May;257(5):863-875. doi: 10.1007/s00417-018-04218-6. Epub 2019 Jan 10. PMID 30627791
- [Background] Calladine D, Evans JR, Shah S, Leyland M. Multifocal versus monofocal intraocular lenses after cataract extraction. Cochrane Database Syst Rev. 2012 Sep 12;(9):CD003169. doi: 10.1002/14651858.CD003169.pub3. PMID 22972061